CLINICAL TRIAL: NCT04540796
Title: A Phase 1, First-in-Human, Dose Escalation Study of the JNJ-75348780 Bispecific Antibody Targeting CD3 and CD22 in Participants With NHL and CLL
Brief Title: A Study of JNJ-75348780 in Participants With Non-Hodgkin Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108882; 75348780LYM1001 (Other: Janssen Research & Development, LLC); 2020-001183-29 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-09-07 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Escalation (Experimental): Participants will receive JNJ-75348780. The dose levels will be escalated sequentially based on the decisions of the Study Evaluation Team (SET), along with the potential exploration of other routes of administration and schedules, until one or more recommended Phase 2 Doses (RP2D) have been identified.
  Interventions: Drug: JNJ-75348780
- Part B: Cohort Expansion (Experimental): Participants will receive JNJ-75348780 at one of the putative RP2Ds determined in Part A.
  Interventions: Drug: JNJ-75348780

INTERVENTIONS:
Drug: JNJ-75348780 — Participants will receive JNJ-75348780 by subcutaneous (SC) administration.

SUMMARY:
The purpose of this study is to characterize safety and to determine the putative recommended Phase 2 dose(s) (RP2D[s]) and optimal dosing schedule(s) of JNJ-75348780 in participants with relapsed/ refractory B-cell Non-Hodgkin Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL) in Part A and to further characterize the safety at the RP2D(s) in Part B.

DETAILED DESCRIPTION:
B-cell lymphoid malignancies include CLL and NHL and are defined by clonal populations of B-lymphocytes expressing identical surface antigens. CD22 is a surface protein specifically expressed on B-lymphocytes and is expressed in B-lymphocytic malignancies. It is known to negatively regulate the B-cell receptor via its cytosolic immunoreceptor tyrosine-based inhibitory motifs. JNJ-75348780 is a novel human bispecific antibody that recognizes the CD3 antigen on T-lymphocytes and the CD22 antigen on mature and malignant B-lymphocytes. JNJ-75348780 is hypothesized to lead to cytotoxicity, T-cell activation, and induction of cytokines upon engagement of CD3 on T-cells and CD22 on malignant B-lymphocytes. The study consists of screening phase, treatment phase and post-treatment phase. The total study duration will be up to 2 years 10 months. Efficacy assessments will include radiographic image assessments, positron emission tomography scan, bone marrow assessment, endoscopy or colonoscopy, physical examinations. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of disease: B-cell NHL or CLL requiring therapy; All participants must have relapsed or refractory disease with no other approved therapies available that would be more appropriate in the investigator's judgment. B cell NHL as defined per the 2016 World Health Organization (WHO) classification: In addition, the following disease-specific criteria outlined below must be met a) If diffuse large B-cell lymphoma (DLBCL): received, or not eligible for high-dose chemotherapy and autologous stem cell transplantation with curative intent, b) If follicular lymphoma (FL)/ marginal zone lymphoma (MZL) (except mucosa-associated lymphoid tissue [MALT]), or Waldenstrom macroglobulinemia (WM): previously treated with a minimum of 2 prior lines of systemic therapy, with at least 1 prior line containing an anti-CD20 antibody, c) If mantle cell lymphoma (MCL): previously treated with at least 1 prior line of systemic therapy containing an anti-CD20 antibody. CLL or small lymphocytic lymphoma (SLL): relapsed or refractory with at least 2 prior lines of therapy to include a bruton tyrosine kinase inhibitor (BTKi) and/or a B-cell lymphoma (BCL)2 inhibitor, if eligible. For Part B: participants must have measurable disease as defined by the appropriate disease response criteria
* Eastern Cooperative Oncology Group (ECOG) performance status Grade of 0 or 1
* Cardiac parameters within the following range: corrected QT interval (QTc intervals corrected using Fridericia's formula [QTcF]) less than or equal to (<=) 480 milliseconds (ms) based on the average of triplicate assessments performed no more than 5 (plus minus [+ -] 3) minutes apart
* Women of childbearing potential must have a negative highly sensitive serum pregnancy test (Beta human chorionic gonadotropin) at screening and prior to the first dose of study drug
* Women must be: a) not of childbearing potential, b) of childbearing potential and practicing a highly effective, preferably user independent method of contraception (failure rate of less than (<) 1 percent (%) per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study drug and until 90 days after last dose

Exclusion Criteria:

* Known central nervous system (CNS) involvement with lymphoma
* Prior solid-organ transplantation
* Either of the following: a) received an autologous stem cell transplant <=3 months before the first dose of JNJ 75348780, b) prior treatment with allogenic stem cell transplant <= 6 months before the first dose of JNJ-75348780, or has evidence of graft versus host disease that requires immunosuppressant therapy
* Prior chemotherapy, targeted therapy, immunotherapy or radiotherapy (with the exclusion of palliative radiation to limited sites that do not interfere with response assessment based on a sufficient number of other sites), within 2 weeks before the first administration of study drug. For investigational agents where the half-life is known, there should be a treatment-free window of at least 2 weeks or 5 half-lives, whichever is longer. For investigational agents with long half-lives a wash-out of 4 weeks is acceptable. Participants who received prior treatment with anti-CD20 * anti-CD3 bispecific therapy will be excluded until a dedicated cohort(s) is opened as determined by the SET
* Active autoimmune disease that requires systemic immunosuppressive medications (example, chronic corticosteroid, methotrexate, or tacrolimus)
* History of malignancy (other than the disease under study in the cohort to which the participant is assigned) within 1 year prior to the first administration of study drug. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy which in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 1 year before the first dose of study drug. Concomitant malignancies that are unlikely to progress and/or preclude evaluation of study endpoints may be allowed after discussion with the Study Responsible Physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 2 years 10 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part A and Part B: Number of Participants with AEs by Severity | Up to 2 years 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Part A and Part B: Number of Participants with Dose-Limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve From Time Zero to End of Dosing Interval (AUCtau) of JNJ-75348780 | Up to 2 years 10 months
  AUCtau is the measure of the serum drug concentration from time zero to end of dosing interval.
Maximum Observed Serum Concentration (Cmax) of JNJ-75348780 | Predose, 48 hours postdose (up to 2 years 10 months)
  Cmax is the maximum observed serum concentration of JNJ-75348780.
Minimum Observed Serum Concentration (Cmin) of JNJ-75348780 | Predose, 48 hours postdose (up to 2 years 10 months)
  Cmin is the minimum observed serum concentration of JNJ-75348780.
Objective Response Rate (ORR) | Up to 2 years 10 months
  ORR is defined as the percentage of participants who achieve a partial response (PR) or better according to the revised response criteria for malignant lymphoma, the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) response criteria and International Workshop for Waldenstrom Macroglobulinemia (IWWM) response criteria.
Complete Response (CR) Rate | Up to 2 years 10 months
  CR rate is defined as the percentage of participants who achieve a best response of CR according to the revised response criteria for malignant lymphoma, iwCLL response criteria and IWWM response criteria.
Time to Response (TTR) | Up to 2 years 10 months
  TTR is defined for participants who achieved PR or CR as the time from the first dose of study drug to first response of PR or CR according to the revised response criteria for malignant lymphoma, iwCLL response criteria and IWWM response criteria.
Duration of Response (DOR) | Up to 2 years 10 months
  DOR is defined for participants who achieved PR or CR as the time between the date of initial documentation of PR or CR to the date of either the first documented evidence of disease progression or death according to the revised response criteria for malignant lymphoma, iwCLL response criteria and IWWM response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (32):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Austin Hospital, Heidelberg
  - Linear Clinical Research Ltd, Nedlands
- France (3):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHU Nantes, Nantes
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
- Israel (5):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky MC, Tel Aviv
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (5):
  - Hospital de Vall D'Hebron, Barcelona
  - Hosp. Univ. Germans Trias I Pujol, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
- Taiwan (5):
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - Leicester Royal Infirmary, Leicester
  - Kings College Hospital, London
  - The Christie Nhs Foundation Trust, Manchester
  - Plymouth Hospital NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency